CLINICAL TRIAL: NCT07226492
Title: A Pilot Trial of an Unconditional Cash Transfer for Pregnant Women With HIV in Botswana
Brief Title: Cash Transfers to Pregnant Women With HIV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: University of Botswana (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 857193; 4K23MH131464-04 (NIH)
Record Dates: First submitted 2025-11-03; First posted 2025-11-10 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: HIV; Pregnancy; HIV Antiretroviral Therapy (ART) Adherence; Post-partum
Keywords: Cash-transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cash-Transfer Intervention (Experimental): Receives usual care and Unconditional Cash Transfers (UCTs) of 1,000 BWP/month
  Interventions: Other: Unconditional Cash Transfer (UCT)
- Usual care (No Intervention): Receives usual care and standard social support

INTERVENTIONS:
Other: Unconditional Cash Transfer (UCT) — Unconditional Cash Transfer (UCT) of 1,000 BWP/month
  Arms: Cash-Transfer Intervention

SUMMARY:
The goal of this study is to evaluate the effectiveness and implementation of an unconditional cash transfer intervention to improve mental bandwidth, ART adherence, and postpartum retention among pregnant women with HIV in Botswana.

The main questions it seeks to answer are:

1. Do unconditional monthly cash transfers improve mental bandwidth relative to usual care among pregnant women with HIV?
2. Do unconditional monthly cash transfers improve ART adherence (PDC) during pregnancy and the postpartum period?
3. Is delivery of UCTs via mobile money feasible and acceptable in public ANC clinics in Botswana?
4. What barriers and facilitators affect implementation, and how should the model be adapted for a larger trial or a policy pilot (e.g., a pregnancy support grant)?

DETAILED DESCRIPTION:
Poverty is an important contributor to poor short- and long-term HIV outcomes for pregnant women with HIV. This problem is salient in Botswana, where antenatal HIV prevalence is >20%. Poverty has been reported as a major barrier to sustained engagement in ART among pregnant women with HIV, and extreme poverty affects 15-20% of people in Botswana. Recent research in behavioral economics has shown that poverty can result in worse health outcomes by taxing mental bandwidth, resulting in a heightened focus on immediate needs and less attention to future-oriented decisions. Mental bandwidth is likely further taxed by the added burdens of HIV and the perinatal period. Consequently, anti-poverty interventions targeting pregnant women with HIV, such as cash transfers, may be particularly effective at improving health outcomes. However, equipoise remains about the role of cash transfers in HIV, with prior studies showing mixed results (e.g., HPTN068 showing no reduction in HIV incidence among school-aged girls receiving cash transfers in South Africa). In addition, there is a policy relevant question of whether and to what extent a pregnancy support grant could help improve outcomes.

In this study, we will conduct a pilot Hybrid Type 2 effectiveness-implementation trial of an unconditional cash transfer intervention for pregnant women with HIV. This research will be conducted at antenatal clinics managed by the District Health Management Teams in Gaborone (e.g., Old Naledi, Mafitlakgosi) and Mogoditsane-Thamaga District (e.g., Lesirane). It will be a collaboration between the University of Botswana and the University of Pennsylvania, through the Botswana-Upenn-Partnership. The study population will be comprised of pregnant women with HIV receiving antenatal care. We will enroll a total of 100 participants in their second trimester - 50 assigned to the usual care arm (standard social support), and 50 assigned to the intervention arm (the addition of 1000 BWP per month through 6 months post partum). All participants will complete study visits at baseline (Visit 1), late pregnancy prior to delivery (Visit 2), and 3-6 months post-partum (Visit 3). Data collected at study visits will include survey questionnaires, bandwidth assessments, and clinical data from the electronic health record database. During the final study visit, we will recruit 20 participants (15 intervention, 5 control; randomly selected) for individual qualitative interviews.

Primary outcomes will include mental bandwidth and ART adherence (effectiveness outcomes), and feasibility and acceptability of the intervention (implementation outcomes). These findings will be used as the basis for an NIH R01 proposal to conduct a larger trial of an unconditional cash transfer powered for clinical outcomes (e.g., postpartum viral suppression).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or greater
* Botswana citizen
* Seeking/receiving antenatal care at antenatal clinics managed by the District Health Management Teams in Gaborone and Mogoditsane-Thamaga District
* Confirmed pregnancy by standard laboratory methods (generally urine testing)
* <20 weeks gestational age (by ultrasound dating)
* HIV seropositive
* Economically vulnerable (self-reported annual income below the Botswana poverty line of 14,000 BWP per year, equivalent to the international poverty line of $2.15 in 2017 purchasing power parity)

Exclusion Criteria:

* Does not meet all of the inclusion criteria
* Unable to provide consent
* Cognitive impairment, per discretion of study staff
* Cannot be in the same household as another enrolled study participant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2028-01-04 (Estimated); Study Completion 2028-01-04 (Estimated)

PRIMARY OUTCOMES:
Antiretroviral Therapy (ART) adherence | From baseline visit through 6 months post-partum
  Proportion of doses covered: Sum of days covered by dispensed medication in the observation period) / (Total number of days in the observation period). This is using pharmacy refill data.
Mental bandwidth: Psychomotor Vigilance Task | At baseline visit, gestational age ≥ 30 weeks (visit 2), 3-6 months post-partum (visit 3)
  Results from Psychomotor Vigilance Task (response time, number of minor lapses and false starts)
Mental bandwidth: Raven's Progressive Matrices | Baseline visit, gestational age ≥30 weeks (visit 2), 3-6 months post-partum (visit 3)
  Raven's Progressive Matrices short form (number of correct answers)
Feasibility of intervention | At gestational age ≥ 30 weeks (visit 2), 3-6 months post-partum (visit 3); qualitative interviews are 3-8 months post-partum
  Feasibility of Intervention Measure, 4-item scale (1-4), higher score indicates greater feasibility; Qualitative interview
Acceptability of intervention | At gestational age ≥ 30 weeks (visit 2), 3-6 months post-partum (visit 3); qualitative interviews are 3-8 months post-partum
  Acceptability of Intervention Measure, 4-item scale (1-4), higher score indicates greater acceptability; Qualitative interview

SECONDARY OUTCOMES:
Food security | At baseline visit, gestational age ≥ 30 weeks (visit 2), 3-6 months post-partum (visit 3)
  Household Hunger Scale - measures the severity of hunger in a household based on experiences of food deprivation over the past 30 days, scale of 1-3, higher number indicates lower food security
Time Preferences (Future Orientation) | At baseline visit, gestational age ≥ 30 weeks (visit 2), 3-6 months post-partum (visit 3)
  Preference Survey Module - measures self-described temporal discounting with a 10-point probabilistic scale; Patience (Brownback) - measures number of weeks willing to wait for an increased payment (delayed economic gratification)
Time Horizon | At baseline visit, gestational age ≥ 30 weeks (visit 2), 3-6 months post-partum (visit 3)
  Time Horizon (Laajaj) - length of time finances are planned in advance
Hope | At baseline visit, gestational age ≥ 30 weeks (visit 2), 3-6 months post-partum (visit 3)
  State Hope Scale, 8-item scale - self-report measure of goal directed thinking, values 1-8, higher value indicates greater hope
Stress | At baseline visit, gestational age ≥ 30 weeks (visit 2), 3-6 months post-partum (visit 3)
  Perceived Stress Scale-4, 5-item scale (assessment of perceived stress over the past 30 days), values 1-5
Psychological Distress | At baseline visit, gestational age ≥ 30 weeks (visit 2), 3-6 months post-partum (visit 3)
  Kessler 6+ (assessment of frequency of psychological distress symptoms over the past 30 days), values 1-5, higher value indicates greater distress
Pregnancy status: pregnant or post-partum | At baseline visit, gestational age ≥ 30 weeks (visit 2), 3-6 months post-partum (visit 3)
  Self-reported status of pregnancy (pregnant or post-partum)
Location of delivery | At 3-6 months post-partum (visit 3)
  Collected from the electronic health record database: whether participant gave birth at a health facility, home, or other
Gestational age at delivery | At 3-6 months post-partum (visit 3)
  Gestational age at delivery, collected from electronic health record database
Birth outcome | 3-6 months post-partum (visit 3)
  Collected from electronic health record database: live birth (child is alive), live birth (child is deceased), still birth, miscarriage, or other
Antenatal HIV clinic attendance | From baseline visit through 6 months post-partum
  From electronic health record database: number of attended visits, number of scheduled visits
Post-partum HIV clinic attendance | From baseline visit through 6 months post-partum
  From electronic health record database: number of attended visits, number of scheduled visits

CONTACTS AND LOCATIONS:
Locations (3):
- Botswana (3):
  - Lesirane Clinc, Gaborone
  - Mafitlhakgosi Clinic, Gaborone
  - Old Naledi Clinic, Gaborone

IPD SHARING:
Plan to Share IPD: No
Sharing IPD is not part of the study's protocol.

REFERENCES:
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Snyder CR, Sympson SC, Ybasco FC, Borders TF, Babyak MA, Higgins RL. Development and validation of the State Hope Scale. J Pers Soc Psychol. 1996 Feb;70(2):321-35. doi: 10.1037//0022-3514.70.2.321. PMID 8636885
- [Background] Laajaj R. Endogenous time horizon and behavioral poverty trap: Theory and evidence from Mozambique. Journal of Development Economics. 2017;127:187-208.
- [Background] Falk A, Becker A, Dohmen T, Huffman D, Sunde U. The Preference Survey Module: A Validated Instrument for Measuring Risk, Time, and Social Preferences. Human Capital and Economic Opportunity Working Group;2016.
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Deitchler M, Ballard T, Swindale A, Coates J. Introducing a simple measure of household hunger for cross-cultural use. Washington, DC: Food and Nutrition Technical Assistance II project, AED. 2011.